CLINICAL TRIAL: NCT02919267
Title: Physiology of Lung Collapse Under One-Lung Ventilation: Underlying Mechanisms
Acronym: PLC-OLV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Jean Bussières, Anesthesiologist, Principal Investigator, Clinical Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IUCPQ 21299
Record Dates: First submitted 2016-09-28; First posted 2016-09-29 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Lung Collapse; One-Lung Ventilation; Thoracic Surgery; Video-Assisted
Keywords: One lung ventilation; Lung collapse; Bronchial blocker; Double lumen tube; video assisted thoracoscopic surgery; VATS; DLT; Thoracic surgery; Video-assisted
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intra-pulmonary pressure determination (Other): A pressure tubing catheter will be connected to the luerlock adaptor of the bronchial blocker (BB) or to the adaptor located on the side of the occluding system mounted at the extremity of the double lumen tube (DLT). The catheter will then be connected to a differential pressure transducer (AD Instruments, Colorado Springs, CO, USA), allowing direct visualisation of the bronchial pressures. Along with intra-bronchial pressure, esophageal pressure will also be measured to eliminate the pressure generated by the positive pressure of the ventilated lung (Adult esophageal balloon catheter, Cooper Surgical, Trumbull, CT, USA). Intra-bronchial pressures will be measured at end-inspiration and end-expiration.
  Interventions: Device: Double lumen tube; Device: Bronchial blocker
- Volume determination (Other): A one-liter bag (Roxon, Etobicoke, ON, Canada) will be filled precisely with 300 mL of air with the use of a calibrated syringe of 3 liters (Hans Rudolph inc, Shawnee, Kansas, United States), through a three-way valve (Hans Rudolph inc, Shawnee, Kansas, United States). Following the filling of the bag, it will be connected to the non-ventilated lumen of the double lumen tube (DLT) or to the bronchial blocker (BB) through the three-way connector. At the end of the observation period, the collector bag will be connected to the calibrated syringe and will emptied from its residual volume.
  Interventions: Device: Double lumen tube; Device: Bronchial blocker

INTERVENTIONS:
Device: Double lumen tube — Either gaseous volume quantification or intrapulmonary pressure measurements will be done in patients randomized in the L-DLT group.
  Other Names: Left-sided double lumen tube (BronchoCath, Mallinkrodt)
Device: Bronchial blocker — Either gaseous volume quantification or intrapulmonary pressure measurements will be done in patients randomized in the BB group.
  Other Names: Bronchial blocker (Fuji Uniblocker, Fuji Systems)

SUMMARY:
Lung isolation technique and one-lung ventilation (OLV) are the mainstays of thoracic anesthesia. Two principal lung isolation techniques are mainly use by clinicians, the double lumen tubes (DLT) and the bronchial blockers (BB). The physiology of lung collapse during OLV is not well described in the literature. Few publications characterized scant aspects of lung collapse, only with the use of DLT and sometime in experimental animals. Two phases of lung collapse have been described. The first phase is a quick and partial secondary to the intrinsic recoil of the lung. The second phase is the reabsorption of gas contained in the alveoli by the capillary bed. The investigators plan to describe the physiology of the second phase of lung deflation using of DLT or BB, in a human clinical context.

DETAILED DESCRIPTION:
Lung isolation and one-lung ventilation (OLV) have been used for more than 60 years, principally via double lumen endotracheal tubes (DLT). Since the beginning of the 21st century, modernisation of bronchial blockers (BB) has favoured their more frequent use. Meanwhile, video assisted thoracoscopic surgery (VATS) has increased, becoming the standard for the majority of intra-thoracic pulmonary surgeries.

Lung collapse during OLV undergoes two distinct phases. The first phase occurs at the opening of the pleural cavity and corresponds to a quick but partial collapse of the lung due to its intrinsic recoil. This phase probably ends when small airways are closed. Thereafter, the second phase, a slower one, corresponds to the reabsorption, by the capillary bed, of gas contained into the alveoli. The speed of this reabsorption depends on the solubility of the gas contained in the alveoli.

Intriguingly, the physiology of lung collapse under OLV remains poorly understood, especially with the use of BB. Theoretically, many aspects of lung isolation may influence lung collapse, including the ventilation strategy before OLV, the timing and the lung isolation devices being used. While oxygen at 100% is widely used for ventilation before OLV, the timing of initiation of lung isolation varies from centers to centers. Indeed, the most conservative will begin the lung isolation just before the opening of the pleural space, whereas others begin the lung isolation following the appropriate positioning of the patient and confirmation that the lung isolation device is properly positioned by fiberoptic bronchoscopy (FOB) examination. Therefore, the period between initiation of lung isolation and pleural opening may vary from a few minutes to >30 minutes. The mechanic of lung isolation differs between DLT and BB and consequently the physiology of lung deflation may be different. When using DLT, the lumen that corresponds to the collapsed lung is disconnected from the ventilator and is continuously in communication with the ambient air. When using BB a bronchial cuff is inflated within the main bronchus following a 30 seconds apnea period, allowing the initial lung deflation to be mediated by elastic lung recoil. After this initial phase, the only communication with ambient air is through the small (2 mm) and long internal (67 mm) channel, which is completely different from the larger lumen of the DLT.

Rapid and complete lung collapse is essential during lung isolation for VATS otherwise; there is no alternative available for the surgeon to get proper view of the pulmonary hilum. Previous studies suggested that BB allow a less effective lung collapse than the one obtained with DLT. However, the authors recently documented that the use of BB with its internal channel occluded creates a statistically significant shorter time to complete lung collapse during VATS compared to DLT (36.6 ± 29.1 vs 7.5 ± 3.8 min; p<0.001). In contrast to the previous studies, the authors used off-line review videos recorded during the surgery to obtain a more objective evaluation of the complete lung collapse time which probably reflected the second phase of lung deflation. Although, our definition of lung collapse was very strict, meaning complete collapse of all the lung areas, graded using a standardized visual scale and chart. However, authors do not have any data to explain why this internal channel occlusion may have some positive impact. The authors hypothesized that their results could be explained by the optimisation of the reabsorption phases following enhanced atelectasis by gas reabsorption (phase 2) after bronchial blockade. This latter hypothesis is supported by a pilot observation that ambient air (FiO2 at 0.21) was "sucked up" within the collapsing lung when using DLT to a greater extent than with the use of BB (unpublished data). The presence of ambient air (21%) in the alveolar space may likely slowing subsequent gas reabsorption compared to intra-alveolar 100% O2 . However, these hypotheses remain to be confirmed.

The investigators proposed this study to update the knowledge about lung collapse with the actual lung isolation devices: DLT and BB. This protocol will describe the lung collapse physiology and allows getting data for the elaboration of further studies.

Thus the present hypothesis is that during the second phase of lung collapse, the inflow of air through the lumen of the non-ventilated lung of the DLT is greater than through the internal channel of the BB, in the course of lung isolation for OLV.

The main objective of this study is the gas volume quantification (GVQ) coming from ambient air towards the alveoli space of the non-ventilated lung during OLV with the use of DLT and BB. These measurements will be performed from the beginning of OLV until 60 minutes after, meaning approximatively 45 minutes after the opening of the pleura by the surgeon. The secondary objective is the intra-pulmonary pressure measurement (IPM) in the non-ventilated lung with the use of DLT and BB during the same period.

ELIGIBILITY:
Inclusion Criteria:

* elective unilateral lung resection (anatomical segmentectomy, lobectomy or pneumonectomy) for lung cancer

Exclusion Criteria:

* anticipated difficult mask ventilation or intubation
* pleural pathology
* previous thoracic surgery
* previous sternotomy
* previous chemotherapy or chest radiotherapy
* severe COPD or asthma (FEV1 ≤ 50%)
* active or chronic pulmonary infection
* endobronchial mass
* tracheostomy

Post randomisation exclusion criteria :

* severe desaturation before or during the observation period
* any clinical situation precluding the use of one of the lung isolation device
* air leak at the level of bronchial isolation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Moreault, MD, Principal Investigator — Laval University; Jean S Bussières, MD, Principal Investigator — Laval University
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Canada

REFERENCES:
- [Background] Shah RD, D'Amico TA. Modern impact of video assisted thoracic surgery. J Thorac Dis. 2014 Oct;6(Suppl 6):S631-6. doi: 10.3978/j.issn.2072-1439.2014.08.02. PMID 25379201
- [Background] Joyce CJ, Baker AB, Kennedy RR. Gas uptake from an unventilated area of lung: computer model of absorption atelectasis. J Appl Physiol (1985). 1993 Mar;74(3):1107-16. doi: 10.1152/jappl.1993.74.3.1107. PMID 8482648
- [Background] Pfitzner J, Peacock MJ, McAleer PT. Gas movement in the nonventilated lung at the onset of single-lung ventilation for video-assisted thoracoscopy. Anaesthesia. 1999 May;54(5):437-43. doi: 10.1046/j.1365-2044.1999.00845.x. PMID 10995140
- [Background] Pfitzner J, Peacock MJ, Harris RJ. Speed of collapse of the non-ventilated lung during single-lung ventilation for thoracoscopic surgery: the effect of transient increases in pleural pressure on the venting of gas from the non-ventilated lung. Anaesthesia. 2001 Oct;56(10):940-6. doi: 10.1046/j.1365-2044.2001.02211.x. PMID 11576095
- [Background] Campos JH, Reasoner DK, Moyers JR. Comparison of a modified double-lumen endotracheal tube with a single-lumen tube with enclosed bronchial blocker. Anesth Analg. 1996 Dec;83(6):1268-72. doi: 10.1097/00000539-199612000-00024. PMID 8942598
- [Background] Bauer C, Winter C, Hentz JG, Ducrocq X, Steib A, Dupeyron JP. Bronchial blocker compared to double-lumen tube for one-lung ventilation during thoracoscopy. Acta Anaesthesiol Scand. 2001 Feb;45(2):250-4. PMID 11167173
- [Background] Campos JH, Kernstine KH. A comparison of a left-sided Broncho-Cath with the torque control blocker univent and the wire-guided blocker. Anesth Analg. 2003 Jan;96(1):283-9, table of contents. doi: 10.1097/00000539-200301000-00056. PMID 12505967
- [Background] Dumans-Nizard V, Liu N, Laloe PA, Fischler M. A comparison of the deflecting-tip bronchial blocker with a wire-guided blocker or left-sided double-lumen tube. J Cardiothorac Vasc Anesth. 2009 Aug;23(4):501-5. doi: 10.1053/j.jvca.2009.02.002. Epub 2009 Apr 10. PMID 19362014
- [Background] Clayton-Smith A, Bennett K, Alston RP, Adams G, Brown G, Hawthorne T, Hu M, Sinclair A, Tan J. A Comparison of the Efficacy and Adverse Effects of Double-Lumen Endobronchial Tubes and Bronchial Blockers in Thoracic Surgery: A Systematic Review and Meta-analysis of Randomized Controlled Trials. J Cardiothorac Vasc Anesth. 2015 Aug;29(4):955-66. doi: 10.1053/j.jvca.2014.11.017. Epub 2014 Dec 2. PMID 25753765
- [Background] Bussieres JS, Somma J, Del Castillo JL, Lemieux J, Conti M, Ugalde PA, Gagne N, Lacasse Y. Bronchial blocker versus left double-lumen endotracheal tube in video-assisted thoracoscopic surgery: a randomized-controlled trial examining time and quality of lung deflation. Can J Anaesth. 2016 Jul;63(7):818-27. doi: 10.1007/s12630-016-0657-3. Epub 2016 May 2. PMID 27138896
- [Background] Merchant R, Chartrand D, Dain S, Dobson J, Kurrek M, LeDez K, Morgan P, Shukla R; Canadian Anesthesiologists' Society. Guidelines to the Practice of Anesthesia Revised Edition 2012. Can J Anaesth. 2012 Jan;59(1):63-102. doi: 10.1007/s12630-011-9609-0. English, French. PMID 22183296
- [Background] Brodsky JB, Lemmens HJ. Tracheal width and left double-lumen tube size: a formula to estimate left-bronchial width. J Clin Anesth. 2005 Jun;17(4):267-70. doi: 10.1016/j.jclinane.2004.07.008. PMID 15950850
- [Background] Fortier G, Cote D, Bergeron C, Bussieres JS. New landmarks improve the positioning of the left Broncho-Cath double-lumen tube-comparison with the classic technique. Can J Anaesth. 2001 Sep;48(8):790-4. doi: 10.1007/BF03016696. PMID 11546721
- [Background] Kovacs G, Avian A, Olschewski A, Olschewski H. Zero reference level for right heart catheterisation. Eur Respir J. 2013 Dec;42(6):1586-94. doi: 10.1183/09031936.00050713. Epub 2013 Jun 21. PMID 23794468
- [Background] Joyce CJ, Baker AB, Parkinson R, Zacharias M. Nitrous oxide and the rate of gas uptake from an unventilated lung in dogs. Br J Anaesth. 1996 Feb;76(2):292-6. doi: 10.1093/bja/76.2.292. PMID 8777113
- [Background] Pfitzner J, Peacock MJ, Pfitzner L. Speed of collapse of the non-ventilated lung during one-lung anaesthesia: the effects of the use of nitrous oxide in sheep. Anaesthesia. 2001 Oct;56(10):933-9. doi: 10.1046/j.1365-2044.2001.02210.x. PMID 11576094
- [Background] Ko R, McRae K, Darling G, Waddell TK, McGlade D, Cheung K, Katz J, Slinger P. The use of air in the inspired gas mixture during two-lung ventilation delays lung collapse during one-lung ventilation. Anesth Analg. 2009 Apr;108(4):1092-6. doi: 10.1213/ane.0b013e318195415f. PMID 19299766
- [Background] Yoshimura T, Ueda K, Kakinuma A, Sawai J, Nakata Y. Bronchial blocker lung collapse technique: nitrous oxide for facilitating lung collapse during one-lung ventilation with a bronchial blocker. Anesth Analg. 2014 Mar;118(3):666-70. doi: 10.1213/ANE.0000000000000106. PMID 24557112
- [Derived] Moreault O, Couture EJ, Provencher S, Somma J, Lohser J, Ugalde PA, Lemieux J, Lellouche F, Bussieres JS. Double-lumen endotracheal tubes and bronchial blockers exhibit similar lung collapse physiology during lung isolation. Can J Anaesth. 2021 Jun;68(6):791-800. doi: 10.1007/s12630-021-01938-y. Epub 2021 Feb 16. PMID 33594596

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As mentioned into the Methods section of the protocol, each patients that were excluded after randomization were replaced by a new randomized patient. We had to randomized 49 patients in order to analyze a total of 39 patients.
Pre-assignment Details: One patient was excluded after the study was completed because when we started the analysis of the results, we realized that one of the patient had an air leak during the study period that was not recognized by the investigator. Since the study was completed, we could not randomized a new patient.
Groups:
- Intra-pulmonary Pressure Measurements With Double-lumen Tube; Intra-pulmonary Pressure Determination With Bronchial Blocker: For patients randomized to the intra-pulmonary pressure measurements, a pressure-tubing catheter was connected to the luerlock adaptor of the BB or to the adaptor located on the side of the occluding system mounted at the extremity of the DLT. The catheter was connected to a differential pressure transducer. Signals were amplified with a CD15 Carrier Demodulator then digitized at 5 Hz and sampled using an MP100 analogic/numeric system. Continuous pressure measurements were recorded before and after pleural opening by the surgeon. Tracings were recorded and subsequent off-line analyses were accomplished using ACQKnowledge and pressures were averaged every 30 seconds, excluding aberrant measures (above and below 2 SD of the mean).
- Gas Movement Quantification With Double-lumen Tube; Gas Movement Quantification With Bronchial Blocker: For patients randomized to the gas movement quantification, a 2-liter bag was filled with 1000 mL of air with a 1000 mL calibrated syringe and a pneumotachometer through a 3-way valve prior to OLV. The pneumotachometer signal was amplified with Pneumotach Amplifier 1 and digitized at 200 Hz using MP100 analogic/numeric system. Volume were measured with ACQKnowledge by integration of flows measured with the pneumotachometer. One minute after initiation of OLV, the three-way valve was connected to the non-ventilated lumen of the DLT or to the internal chanel of the BB through an adaptor. Immediately prior to opening of the pleura, the volume measurement bag was closed and apnea was re-established in both groups for one minute as described above, after which measurements resumed for a total duration of 60 minutes of OLV. At the end of the observation period, the bag was emptied with the one-liter syringe through the pneumotachometer to measure its residual volume.
Period: Overall Study
Arm/Group | Intra-pulmonary Pressure Measurements With Double-lumen Tube | Intra-pulmonary Pressure Determination With Bronchial Blocker | Gas Movement Quantification With Double-lumen Tube | Gas Movement Quantification With Bronchial Blocker
Started | 10 | 12 | 13 | 14
Completed | 10 | 9 | 10 | 10
Not Completed | 0 | 3 | 3 | 4
Not completed — Protocol Violation | 0 | 3 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intra-pulmonary Pressure Measurements With Double-lumen Tube | Intra-pulmonary Pressure Determination With Bronchial Blocker | Gas Movement Quantification With Double-lumen Tube | Gas Movement Quantification With Bronchial Blocker | Total
Number analyzed (Participants) | 10 | 9 | 10 | 10 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10) | 67 (7) | 64 (13) | 64 (13) | 63 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 8 | 7 | 28
  Male | 3 | 3 | 2 | 3 | 11
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 73 (21) | 76 (26) | 66 (12) | 65 (10) | 70 (18)
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 163 (7) | 163 (10) | 160 (10) | 162 (12) | 162 (10)
BMI (kg/m2) [Mean (Standard Deviation); unit: kilograms/m^2] | 28 (8) | 28 (7) | 26 (5) | 25 (4) | 27 (6)
Forced expiratory volume in one second (FEV1) (% of predicted) [Mean (Standard Deviation); unit: % of predicted value] | 86 (21) | 90 (14) | 92 (20) | 93 (20) | 90 (18)
Time tu pleural opening (min) [Mean (Standard Deviation); unit: minutes] | 14 (6) | 12 (6) | 12 (4) | 14 (4) | 13 (5)
Side of surgery (R/L) [Count of Participants; unit: Participants] — Side of surgery (right vs left)
  Participants
    Right-sided surgery | 7 | 6 | 6 | 5 | 24
    Left-sided surgery | 3 | 3 | 4 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Quantification of Gas Volume Coming From Ambient Air Towards the Alveoli Space of the Non-ventilated Lung During OLV With the Use of DLT and BB.
Time Frame: From the beginning of OLV until 60 minutes
Measure: Mean (Standard Error); unit: milliliters (mL)
Arm/Group | Gas Movement Quantification With Double-lumen Tube | Gas Movement Quantification With Bronchial Blocker
Number analyzed (Participants) | 10 | 10
milliliters (mL) | 504 (85) | 630 (86)

2. Secondary Outcome: Measurement of Intra-pulmonary Pressure in the Non-ventilated Lung With the Use of DLT and BB
Description: Intra-pulmonary pressure measured from initiation of OLV to pleural opening were similarly analyzed using a two-way ANOVA. Two experimental factors, one associated to the comparison between two groups (DLT versus BB), factor fixed and one associated to the comparison among results from the time periods (0 to 10 minutes), factor fixed with interaction terms between the fixed factors were defined. The data was analyzed using a repeated mixed model. An autoregressive covariance structure was used to consider the dependency among repeated measurements.
Time Frame: From the beginning until 10 minutes of OLV
Measure: Mean (Standard Error); unit: cmH2O
Arm/Group | Intra-pulmonary Pressure Measurements With Double-lumen Tube | Intra-pulmonary Pressure Determination With Bronchial Blocker
Number analyzed (Participants) | 9 | 10
cmH2O
  0 minutes | 0 (0) | 0 (0)
  1 minutes | -1.1 (0.3) | -0.7 (1.2)
  2 minutes | -2.4 (0.4) | -2.6 (1.7)
  3 minutes | -3.7 (0.6) | -4.9 (2.6)
  4 minutes | -5.2 (0.9) | -8.9 (4.5)
  5 minutes | -6.9 (1.3) | -11.9 (5.6)
  6 minutes | -8.8 (1.8) | -14.2 (8)
  7 minutes | -10.7 (2.3) | -18.1 (9.4)
  8 minutes | -13.6 (3.1) | -19.7 (9.2)
  9 minutes | -16.3 (3.8) | -24.6 (12.0)
  10 minutes | -20.6 (4.9) | -28.3 (13.6)

ADVERSE EVENTS:
Arm/Group | Intra-pulmonary Pressure Measurements With Double-lumen Tube | Intra-pulmonary Pressure Determination With Bronchial Blocker | Gas Movement Quantification With Double-lumen Tube | Gas Movement Quantification With Bronchial Blocker
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12 | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/13 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No